CLINICAL TRIAL: NCT04601766
Title: A Phase I, Open-Label, Randomized, Two-phase, Crossover Study to Evaluate the Safety, Tolerability and Pharmacokinetics of APL-1501 ER Tablets 2, APL1501 ER Tablets 3, and APL-1202 in Healthy Volunteers
Brief Title: A Phase I, Two-phase, Crossover Study to Evaluate the Safety, Tolerability and Pharmacokinetics of APL-1501 ER Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asieris Pharmaceuticals (AUS) Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHGT-PN-01
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2020-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: APL-1202+APL-1501 ER Tablets 3+APL-1501 ER Tablets 2
- Group B (Experimental)
  Interventions: Drug: APL-1501 ER Tablets 3+APL-1202+APL-1501 ER Tablets 2

INTERVENTIONS:
Drug: APL-1202+APL-1501 ER Tablets 3+APL-1501 ER Tablets 2 — Phase1: Period 1 drug administration( APL-1202 50 mg, 3 tablets, orally );Washout( 7± 1 day) ; Period 2 drug administration(1501 ER Tablets 3 382 mg ASN-1324, 1 tablet); Phase2:Washout(The initiation of second phase will depend on the results of first phase within 30 days and not less than 7 days after the first phase ); Period 3 (APL-1501 ER Tablets 2,382 mg ASN-1324, 1 tablet)
  Arms: Group A
Drug: APL-1501 ER Tablets 3+APL-1202+APL-1501 ER Tablets 2 — Phase1: Period 1 drug administration( 1501 ER Tablets 3 382 mg ASN-1324, 1 tablet );Washout( 7± 1 day) ; Period 2 drug administration(APL-1202 50 mg, 3 tablets, orally); Phase2:Washout(The initiation of second phase will depend on the results of first phase within 30 days and not less than 7 days after the first phase ); Period 3 (APL-1501 ER Tablets 2,382 mg ASN-1324, 1 tablet)
  Arms: Group B

SUMMARY:
A two-phase study design will be used for this pilot study. In the first phase, a 2×2 crossover study will be used to evaluate the safety, tolerability and PK characteristic of APL-1202 and APL-1501 ER Tablets 3. Twelve healthy subjects will be in ratio 1:1 randomly assigned to two groups, randomization will be stratified by gender (male, female) in ratio 1:1. Each group will be dosed with APL-1202, APL-1501 ER Tablets 3 in a cross-over way. A 7-day (±1 day) washout will be required before next period of drug administration. The samples in first phase will be sent to bioanalysis lab for PK research at the end of first phase. The initiate of second phase will depend on the results of first phase within 30 days and not less than 7 days after the first phase.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have informed consent before the trial, and have a full understanding of the content, process and possible adverse reactions of the trial, and voluntarily signed a written informed consent form
2. The subject is able to communicate well with the researchers and is able to complete the trial in accordance with the protocol
3. 18 to 45 years old (including 18 and 45 years old)
4. Postmenopausal females or sterilized participant must be at least 6 months post-menopausal, surgically sterile; the postmenopausal/sterilization should be confirmed by FSH testing
5. The body weight of male subjects are ≥ 50 kg, and that of female subjects are ≥ 45 kg, and the body mass index (BMI) are between 18.0 and 30.0 kg/m2, including the boundary value. BMI= weight (kg) / height2 (m2)
6. Must have normal organ functions, including the following:

   1. Bone marrow reserve: within normal range or deemed NCS by the treating investigator
   2. Hepatic: total bilirubin within normal range or deemed NCS by the treating investigator; aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 1.5x ULN
   3. Renal: serum creatinine ≤ ULN Confidential Page 7 of 61
   4. Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ ULN or deemed NCS by the treating investigator
   5. QTCF≤450 msec for males and 470 msec for females
7. Healthy as determined by physician, based on a medical evaluation including Physical examination and vital signs, hematology, biochemistry, coagulation, urinalysis, and 12-lead Electrocardiograms (ECGs)
8. Willingness for subjects of reproductive potential to use highly effective methods of contraception from the beginning of the study screening to the end of study follow up period a. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year, when used consistently and correctly)

Exclusion Criteria:

1. History of allergy to any research drug components, similar drugs or their excipients
2. History of optic nerve disorder, malignancy, anemia or gastrointestinal, liver and kidney diseases that may affect the pharmacokinetics of the investigational drugs
3. Subject who is positive in one or more of the tests of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), and AIDS antibody (HIV)
4. Subject who is positive for urine drug screening or who with a history of drug abuse
5. Subject who smoked more than 5 cigarettes per day in the 3 months before the trial, and/or disagreed to avoid using any tobacco products 24 hours before administration and during hospitalization
6. Regular drinkers within 6 months before the trial, that is, those who drank more than 14 units of alcohol per week (1 unit = 10 g pure alcohol), and/or those who do not agree to stop alcohol intake 24 hours before administration and during hospitalization, and/or positive in breath alcohol test. STANDARD DRINK= Volume of Alcoholic Drinks x Concentration of Alcoholic Drinks x 0.789/pure alcohol
7. Systemic treatment on any investigational clinical trial within 28 days (or 5 half-lives of that agent, whichever is greater) prior to enrollment
8. Subject who take strong inducers or inhibitors of metabolism enzymes or transporter within 48 h before the study, including but not limited to caffeine, xanthine, grapefruit, grapefruit juice or grapefruit-related citrus fruits (e.g. Seville oranges, pomelos) etc.
9. Pregnancy or lactation
10. Any other reason that in the opinion of the Investigator or Sponsor would prevent the patient from completing participation or following the study schedule

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
AEs | 6 months
  Number of subjects with AEs,
SAEs | 6 months
  Number of subjects with SAEs

SECONDARY OUTCOMES:
PK parameters: area under the curve (AUC) | 6 months
  Area under the curve (AUC) of APL-1501 ER Tablets, and APL-1202 Tablets
PK parameters: maximum concentration (Cmax) | 6 months
  maximum concentration (Cmax), of APL-1501 ER Tablets, and APL-1202 Tablets
PK parameters: Tmax | 6 months
  Tmax of APL-1501 ER Tablets, and APL-1202 Tablets
PK parameters: half-life | 6 months
  apparent t1/2 of APL-1501 ER Tablets, and APL-1202 Tablets
Urine concentration | 6 months
  Urine concentration of APL-1501 ER Tablets 2, APL-1501 ER Tablets 3, and APL-1202 Tablets.
Accumulated excretion rate (Ae%) | 6 months
  Accumulated excretion rate (Ae%) of APL-1501 ER Tablets 2, APL-1501 ER Tablets 3, and APL-1202 Tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia clinical research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No